CLINICAL TRIAL: NCT01775761
Title: A Randomized, Placebo- And Positive-Controlled Cross-Over Study To Evaluate The Effect Of Tafamidis On The QTC Interval In Healthy Volunteers
Brief Title: A Study To Determine Any Effect Of Tafamidis On Electrocardiographic Intervals, Specifically The Rate Corrected QT Interval (QTc)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: B3461031
Record Dates: First submitted 2013-01-15; First posted 2013-01-25 (Estimated); Last update posted 2013-05-21 (Estimated); Status verified 2013-05

CONDITIONS: TTR Cardiomyopathy
Keywords: Thorough QTc evaluation of tafamidis compared to the effects of moxifloxacin and placebo in healthy volunteers.
MeSH Terms: interventions — tafamidis; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- Period 1: 960 mg tafamidis (Vyndaqel) (Experimental)
  Interventions: Drug: Period 1
- Period 2: 400 mg moxifloxacin (Experimental): 400 mg moxifloxacin
  Interventions: Drug: Period 2
- Period 3: Placebo (Experimental)
  Interventions: Drug: Period 3

INTERVENTIONS:
Drug: Period 1 — A comparison of less than or equal to 960 mg tafamidis, 400 mg moxifloxacin and placebo on the rate corrected QT interval.
  Other Names: tafamidis (Vyndaqel)
  Arms: Period 1: 960 mg tafamidis (Vyndaqel)
Drug: Period 2 — A comparison of less than or equal to 960 mg tafamidis, 400 mg moxifloxacin and placebo on the rate corrected QT interval.
  Other Names: moxifloxacin
  Arms: Period 2: 400 mg moxifloxacin
Drug: Period 3 — A comparison of less than or equal to 960 mg tafamidis, 400 mg moxifloxacin and placebo on the rate corrected QT interval.
  Arms: Period 3: Placebo

SUMMARY:
The purpose of this study is to investigate the effects of tafamidis on the intervals of the electrocardiogram, specifically the rate corrected QT interval (QTc) in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, nonsmoking, male and/or female subjects of non-childbearing potential.
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2.
* Total body weight >50 kg (110 lbs).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease.
* An ALT or AST measurement >2 times the ULN.
* 12-lead ECG demonstrating QTc >450 msec or a QRS interval >120 msec at Screening.
* Subjects at increased risk if dosed with moxifloxacin, according to the product label for moxifloxacin.
* History of risk factors of QT prolongation or torsades de pointes, congenital deafness and family history of sudden death.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2013-01; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
QTc interval using Fridericia's correction method (QTcF) of tafamidis and placebo (baseline-adjusted) at each post-dose time | SCRN, -1, -0.5, 0, 1, 1.5, 2, 3, 4, 6, 12, 24 hrs

SECONDARY OUTCOMES:
QTcF of moxifloxacin and placebo at historical moxifloxacin median Tmax of 3 hours. | Scrn, -1, -0.5, 0, 1, .5, 2, 3, 4, 6, 8, 12, 24 hrs
Tmax | 0, 1, .5, 2, 3, 4, 6, 8, 12, 24 hrs
Cmax | 0, 1, .5, 2, 3, 4, 6, 8, 12, 24 hrs
AUC0-24 | 0, 1, .5, 2, 3, 4, 6, 8, 12, 24 hrs

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- Pfizer Investigational Site, New Haven, Connecticut, United States
- Pfizer Investigational Site, Brussels, Belgium
- Pfizer Investigational Site, Singapore, Singapore, Singapore

REFERENCES:
- [Derived] Klamerus KJ, Watsky E, Moller R, Wang R, Riley S. The effect of tafamidis on the QTc interval in healthy subjects. Br J Clin Pharmacol. 2015 Jun;79(6):918-25. doi: 10.1111/bcp.12561. PMID 25546001
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B3461031&StudyName=A%20Study%20To%20Determine%20Any%20Effect%20Of%20Tafamidis%20On%20Electrocardiographic%20Intervals%2C%20Specifically%20The%20Rate%20Corrected%20QT%20Interval%20%28QTc%29